CLINICAL TRIAL: NCT06253364
Title: A Robust Biomarker of Aggressive HCC and the Response for Adjuvant PD-1 Inhibitors or Combined TKIs Following Liver Resection: Vessels That Encapsulate Tumor Clusters
Brief Title: VETC is an Effective Marker for Postoperative Adjuvant Immunotherapy
Status: Completed | Type: Observational
Sponsor: Chen Xiaoping (Other)
Responsible Party: Sponsor-Investigator, Chen Xiaoping, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: Biomarker1
Record Dates: First submitted 2024-02-03; First posted 2024-02-12 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: HCC; Recurrence
MeSH Terms: conditions — Recurrence | interventions — lenvatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Liver resection group: No adjuvant therapy after hepatectomy.
- Adjuvant PD-1 group: Adjuvant therapy with PD-1 monoclonal antibody after hepatectomy
  Interventions: Drug: PD-1 monoclonal antibody and lenvatinib
- Adjuvant PD-1 plus Lenvatinib group: Adjuvant therapy with PD-1 monoclonal antibody combined with lenvatinib after hepatectomy.
  Interventions: Drug: PD-1 monoclonal antibody and lenvatinib

INTERVENTIONS:
Drug: PD-1 monoclonal antibody and lenvatinib — Adjuvant PD-1 group: Patient receives first adjuvant PD-1 monoclonal antibody 2-4 weeks postoperatively, 200mg IV over 21 days for 9 cycles.
  Adjuvant PD-1 plus Lenvatinib group: Patient receives first adjuvant PD-1 monoclonal antibody 2-4 weeks postoperatively, 200 mg IV 21 days for 9 cycles; lenvatinib is initiated orally 2-4 weeks postoperatively for 6 months.
  Groups: Adjuvant PD-1 group; Adjuvant PD-1 plus Lenvatinib group

SUMMARY:
Vessels that encapsulate tumor clusters (VETC) is an invasive metastatic factor in HCC independent of the epithelial mesenchyme transition (EMT), and VETC-positive patients have a higher rate of postoperative recurrence. However, it is not clear how the surgical prognosis of VETC-positive patients can be improved.

DETAILED DESCRIPTION:
Previous studies have identified VETC as a new metastatic pattern independent of EMT that may be associated with immunosuppression as well as poor prognosis. Multiple retrospective studies find higher rates of postoperative recurrence, distant metastasis in VETC-positive patients. How to improve surgical prognosis in VETC-positive patients needs to be explored. There is no consensus on postoperative adjuvant therapy for HCC. In recent years, adjuvant immunotherapy (sintilimab) and adjuvant immunotherapy combined with targeted therapy (T+A) have been shown to be effective in improving the surgical prognosis. Therefore, the investigators retrospectively collected three surgical resection cohorts, the surgical resection alone group, the postoperative adjuvant PD-1 monotherapy group, and the postoperative adjuvant PD-1 monotherapy combined with Lenvatinib group, to compare these postoperative adjuvant therapies in a subgroup of VETC patients.

ELIGIBILITY:
Inclusion Criteria:

* Underwent radical hepatectomy
* No preoperative treatment
* Pathological confirmed HCC
* High-risk recurrent HCC
* Not receiving any adjuvant therapy or receiving adjuvant therapy with PD-1 monotherapy or receiving adjuvant therapy with PD-1 monotherapy in combination with Lenvatinib after surgery

Exclusion Criteria:

* Macrovascular invasion
* No available wax blocks
* No complete clinical information

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who met the inclusion and exclusion criteria were retrospectively collected for this study.
Sampling Method: Non-Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Disease -free survival | From date of include in this research until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 60 months
  Disease-free survival was defined as defined as the time from enrollment to diagnosis of recurrence or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No